CLINICAL TRIAL: NCT02560675
Title: Why Does Acute Post Whiplash Injury Pain Transform Into Chronic Pain? Multi-modal Assessment of Risk Factors and Predictors of Pain Chronification
Brief Title: Why Does Acute Post Whiplash Injury Pain Transform Into Chronic Pain?
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 601-14-RMB Whiplash_CTIL; 597-14-RMB Gene_Whiplash_CTIL (Other: Rambam Genetic sub study)
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain Due to Injury
Keywords: Whiplash Injury Pain; Chronic Pain; TBI
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection for genetics. Whole blood sample (10cc) will be collected from each subject and placed in EDTA-coated tubes. Genomic DNA will be isolated using DNA Extraction Kit . Quality and quantity of the DNA sample will be measured using a NanoDrop Machine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 120 healthy subjects: One hundred and twenty healthy subjects (range 20-79; 20 subjects per age decade, 10 M and 10 F) will participate in the first phase of the study aimed to collect normative data from healthy population.
  Study design Phase I - Normative data collection for the inhibitory and excitatory pain modulation responses, a study on healthy subjects (no blood tests)
- 750 subjects with acute whiplash-injury: Seven hundred and fifty acute whiplash-injury based mild TBI will participate in this study.
  Phase II - Multi-modal assessment of acute mild TBI whiplash patients and follow-up

SUMMARY:
Why does acute post whiplash injury pain transform into chronic pain? Multi-modal assessment of risk factors and predictors of pain chronification

DETAILED DESCRIPTION:
Background

The proposed study aims to explore why acute pain turns, in some patients, into chronic pain, and to develop tools for prediction of this transition. Based on the clinical and psychological assessment along with psychophysical and neurophysiological assessment of pain perception, with the analysis of connectivity between several brain centers relevant for pain processing, together with pain genetics, we expect to develop a tool, that will predict, for the individual patient with acute pain inflicted by a whiplash injury, what are the chances for him/her to go into chronic pain situation. Further, by knowing the dysfunctions of pain processing that a patient has, it will be possible to offer the treatment of highest chances to succeed.

Our specific aims are to evaluate, in the setup of acute whiplash injury, the risk of transition to chronic pain based on each of the following testing domains: (i) Psychophysical and neurophysiological data describing facilitatory and inhibitory modulation capacity of the patient. (ii) Psychological data describing patient's behavior such as catastrophizing, fear of pain, post-traumatic stress and depressed mood. (iii) Structural and functional neuro-imaging data describing brain anatomy and function, where we assess resting state MRI activity, grey matter properties using T1 weighted imaging, and white matter properties using diffusion tensor imaging. (iv) Genetic data describing the genetic epidemiology of every patient for the examination of genetic variants associated with transition to chronic pain, and (v) individual case data related to age, gender, education, socioeconomic parameters and personal medical history, as well as features of the specific injury. Overall, we aim to construct a composite scoring system, based on the most relevant of the above mentioned parameters, yielding the highest relative predictive value in identifying acute pain patients who have higher risk for chronification.

Subjects One hundred and twenty healthy subjects (range 20-79; 20 subjects per age decade, 10 M and 10 F) will participate in the first phase of the study aimed to collect normative data from healthy population.

Seven hundred and fifty acute whiplash-injury based mild traumatic brain injuries (TBI) will participate in this study.

Study design Phase I - Normative data collection for the inhibitory and excitatory pain modulation responses, a study on healthy subjects

Phase II - Multi-modal assessment of acute mild TBI whiplash patients and follow-up

1. Initial experimental assessment, will consist, in most cases, of two sessions, one during the ER visit, and the next within 72 hrs of injury, pending on team and device availability, such that all tests will be completed, as follows:

   1. Physical examination with a full neurological exam, and assessment of neck movement.
   2. Psychophysical pain measurements:

   i. Pain thresholds. ii. Suprathreshold pain magnitude estimation; iii. Mechanical temporal summation (TS) and electrical TS iv. Conditioned pain modulation (CPM) - as described for the phase I protocol. It is noted that similar protocols of pain measurement are commonly performed in many labs worldwide in many acute and chronic pain setups, and are considered safe, with no damaging effect on the disease state.

   c. Psychological examination via filling questionnaires for evaluation the following variables: i. Pain Catastrophizing ii. Depression iii. Post-traumatic Diagnostic Scale (PDS) iv. Fear of pain v. The perceived stress of the subjects is assessed by the validated Hebrew version Cohen's Perceived Stress Scale (PSS).

   vi. Five factor model (FFM)

   d.Blood collection for genetics. Whole blood sample (10cc) will be collected from each subject and placed in Ethylenediaminetetraacetic acid (EDTA)-coated tubes. Genomic DNA will be isolated using DNA Extraction Kit . Quality and quantity of the DNA sample will be measured using a NanoDrop Machine.

   e. Magnetic resonance imaging (MRI)/Functional MRI (fMRI) examination in a 3T scanner.

   f. Neurophysiological assessment of pain modulation with 64-channel EEG recording (Brain Products GmbH, Munich, Germany) of CPM and TS.

   i.Neurophysiological assessment of CPM ii.Neurophysiological assessment of TS will be based on electrical evoked potentials obtained with a constant current stimulator
2. Follow up Patients will self-report their pain levels and use of analgesics once in two weeks.

At 6 and 12 month visits patients will be invited to repeat the psychophysical and neurophysiological pain assessments and psychological questionnaires. Selected patients will undergo a second MRI assessment.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of whiplash injured in road accident up to 72h before ER arrival; Glasgow coma scale 13-15 and no traumatic brain findings in computed tomography (CT); no, or shorter than 30 minutes loss of consciousness in the accident. Age 18-70, both males and females.

Exclusion criteria:

Other major bodily injuries at present accident; intracranial hemorrhage or skull fracture in present accident, prior chronic head/neck pain that requires treatment on regular basis; neurological disease that might affect performance of the tests or their interpretation such as neurodegenerative diseases; head and neck injury in past year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 750 Subjects with acute post whiplash injury pain. and 120 healthy subjects .
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Chronic pain | 12 months
  acute post whiplash injury pain transform into chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Principal Investigator — Head of Neurology department at Rambam
Locations (1):
- Rambam Health Care Campus, Haifa, Israel